CLINICAL TRIAL: NCT03752268
Title: Development of an Intervention to Enhance Cancer Pain Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Lara Traeger, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 13-614; ACS MRSG 14-107-01 (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Other Cancer
Keywords: Other Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhancing Cancer Pain Management Part 1 (No Intervention): * Will collect information from participants via self-report assessment at two time points: at baseline (i.e. study enrollment) and approximately 8 weeks post-baseline
  * Will then use MEMS to monitor LA opioid intake over approximately 8 weeks
  * A subset of enrolled participants (n=20) will be invited to participate in an optional one-time qualitative exit interview with a study staff member trained in conducting qualitative interviews
- Enhancing Cancer Pain Management Part 2 (Experimental): * Enhancing Cancer Pain Management will consist of 3 individual manualized sessions
  * The 3 individual manualized sessions will be conducted (approximately 20 minutes each), led by a nurse practitioner, to provide sufficient dose for change in adherence behaviors.
  * Learning and practicing skills for managing cancer-related pain and adhering to prescribed LA opioid regimens.
  * Study staff will provide participants with MEMS caps and bottles at time of enrollment, to monitor LA opioid intake over approximately 14 weeks.
  Interventions: Behavioral: Enhancing Cancer Pain Management

INTERVENTIONS:
Behavioral: Enhancing Cancer Pain Management — Patients will learn and practice an enduring framework of cognitive-behavioral strategies, to enhance adherence behavior, reduce intentional and unintentional deviations from the prescribed regimen.
  Arms: Enhancing Cancer Pain Management Part 2

SUMMARY:
This research study is being done to understand how patients with chronic cancer pain take their long-acting opioid medications, and to develop an intervention to enhance cancer pain management.

DETAILED DESCRIPTION:
Long-acting opioids are a common treatment for cancer pain. The purpose of this study is to develop a program for patients who are taking a prescribed long-acting opioid for their cancer pain. Participants will be enrolled in this study at the Massachusetts General Hospital Cancer Center. This 14-week study involves completing a set of questionnaires at three different times during the study period. . During the study period, participants will use electronic pill caps to monitor their pain medication taking. They also will attend a series of three visits with one of the nurse practitioners on their care cancer team. The visits will focus on learning and practicing skills for managing cancer pain. The information that the investigators collect will help identify whether the sessions are feasible and useful to patients during the course of treatment for cancer pain.

This trial will consist of two parts:

Part 1: This is a single-group prospective observational study. Investigators will use quantitative and qualitative methods to examine rates, predictors and outcomes of adherence to LA opioids over a period of approximately eight weeks. This information will be used to inform Part 2 intervention development and testing.

Part 2: Investigators will test the behavioral intervention in a non-randomized open pilot, over a period of approximately six weeks. Intervention process data, psychosocial and medical data, and post-intervention feedback will be collected to assess feasibility and acceptability. In an iterative process, ongoing data from exit interviews and therapist experience will be used to modify the intervention protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or older
* Currently prescribed a long-acting (LA) opioid for nociceptive cancer pain (extended release oxycodone, extended-release morphine, transdermal fentanyl patches, methadone tablets)
* Ability to comprehend study materials in English
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* In charge of administering own pain medications
* Part 2 study only: within 4 months of current prescription of LA opioid for nociceptive cancer pain

Exclusion Criteria:

* Impaired cognition, active substance disorder, or other active, unstable mental health disorder
* Current long-acting opioid treatment for pre-existing condition
* Part 2 study only: Prior enrollment in the Part 1 study**

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-04-15 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who complete study sessions | 2 Years
  Proportion of enrolled participants who complete the study, based on a criterion of greater than or equal to 75% completed sessions.
Number of participants who identify study components as acceptable | 2 years
  Individual response frequencies of 4 Likert-type scale items, designed for this study, that rate acceptability of 1) number of study sessions, 2) length of study sessions, 3) usefulness of study material, and 4) impact of study material on pain management, and themes of two free-text items that elicit unstructured participant feedback about acceptability of these study components.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Traeger, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No